CLINICAL TRIAL: NCT06775743
Title: ORIENT-31 Regimen (Sintilimab Plus Bevacizumab Plus Platinum-doublet Chemotherapy) in Combination with Stereotactic Radiotherapy in EGFR-mutant Metastatic Non-small Cell Lung Cancer After First-line Third-generation EGFR Tyrosine Kinase Inhibitors (ORBIT Study)
Brief Title: ORIENT-31 Regimen in Combination with SBRT for EGFR-mutant Metastatic NSCLC After First-line Third-generation EGFR-TKIs
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhengfei Zhu, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORBIT
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2025-01

CONDITIONS: NSCLC (advanced Non-small Cell Lung Cancer); EGFR Mutation Positive Advanced Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SBRT plus ORIENT-31 regimen (Experimental)
  Interventions: Drug: ORIENT-31 regimen; Radiation: SBRT

INTERVENTIONS:
Drug: ORIENT-31 regimen — Sintilimab plus bevacizumab plus platinum-doublet chemotherapy
Radiation: SBRT — Based on the results of the response evaluation, personalized SBRT will be arranged after cycle 4:
  A. Complete response, CR: continue with maintenance therapy of PD-1 antibody + pemetrexed + VEGF antibody until disease progression, intolerable toxic side effects, or up to two years.
  B. Stable disease, SD/partial response, PR: if the residual lesions do not exceed three organs and five lesions, and if the investigator deems SBRT feasible, curative-dose stereotactic radiotherapy covering all residual lesions will be administered, with dosing based on the NRG-BR001 study.
  C. If the residual lesions exceed three organs or five lesions, SBRT (24 Gy/3 Fx) targeting 1-3 selected tumor lesions will be performed, and then continue with maintenance therapy of PD-1 antibody + pemetrexed + VEGF antibody until disease progression.
  D. Progressive disease, PD: subsequent treatment is conducted according to the standard guidelines.

SUMMARY:
The goal of this prospective study is to explore the safety and preliminary efficacy of stereotactic body radiotherapy (SBRT) combined with ORIENT-31 regimen (Sintilimab plus bevacizumab plus platinum-doublet chemotherapy) for advanced epidermal growth factor receptor (EGFR)-mutated non-small cell lung cancer (NSCLC) patients who failed first-line third-generation epidermal growth factor receptor-tyrosine kinase inhibitor (EGFR-TKI) treatment. Participants will first receive the standard four-drug combination therapy: PD-1 antibody + vascular endothelial growth factor (VEGF) antibody + platinum + pemetrexed. The efficacy will be evaluated every two courses. According to the efficacy evaluation results, personalized SBRT was be administered.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status score of 0-1;
* Histologically or cytologically confirmed stage IV primary non-small cell lung cancer;
* EGFR-sensitive mutations (L858R, 19del);
* Resistance to first-line treatment with third-generation EGFR-TKIs;
* At least one measurable lesion;
* Patients with brain metastases may be included, but they must be asymptomatic neurologically and have stable lesions without the need for systemic corticosteroid treatment;
* Men and women of reproductive age agree to contraception during the trial (surgical sterilization or oral contraceptives/intrauterine device + condoms);
* Life expectancy ≥ 3 months;
* Within one week before enrollment, organ function levels must meet the following criteria:

  1. Bone marrow function: Hemoglobin ≥ 80 g/L, white blood cell count ≥ 4.0 × 10^9/L or neutrophil count ≥ 1.5 × 10^9/L, platelet count ≥ 100 × 10^9/L;
  2. Liver: Serum total bilirubin level ≤ 1.5 times the upper limit of normal, and when serum total bilirubin level > 1.5 times the upper limit of normal, direct bilirubin level must be ≤ the upper limit of normal, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times the upper limit of normal;
  3. Kidney: Serum creatinine level < 1.5 times the upper limit of normal or creatinine clearance rate ≥ 50 ml/min, blood urea nitrogen ≤ 200 mg/L; serum albumin ≥ 30 g/L;
* Patients must have the capacity to understand and voluntarily sign the informed consent form.

Exclusion Criteria:

* Patients with severe autoimmune diseases: active inflammatory bowel disease (including Crohn's disease, ulcerative colitis), rheumatoid arthritis, scleroderma, systemic lupus erythematosus, autoimmune vasculitis (such as Wegener's granulomatosis), etc.
* Symptomatic interstitial lung disease or active infectious/non-infectious pneumonia.
* Patients with risk factors for intestinal perforation: active diverticulitis, intra-abdominal abscess, gastrointestinal (GI) obstruction, abdominal cancer, or other known risk factors for intestinal perforation.
* History of other malignant tumors.
* Patients with active infections, heart failure, myocardial infarction within the past 6 months, unstable angina, or unstable arrhythmias.
* Physical examination or clinical laboratory findings that the investigator believes may interfere with the results or increase the risk of treatment complications, or other uncontrollable diseases.
* Patients whom the investigator believes currently have lesions requiring palliative radiation therapy.
* Mixed with small cell lung cancer components.
* Nursing or pregnant women.
* Congenital or acquired immunodeficiency diseases including human immunodeficiency virus (HIV), or history of organ transplantation or allogeneic stem cell transplantation.
* Known hepatitis B virus (HBV), hepatitis C virus (HCV), or active tuberculosis infection.
* Patients who have received cancer vaccines or received other vaccines within 4 weeks before starting treatment (Note: Seasonal influenza vaccines are often inactivated vaccines and are allowed, while intranasal preparations are usually live attenuated vaccines and are not allowed).
* Patients who are concurrently using other immunotherapies, chemotherapy drugs, drugs from other clinical trials, or require long-term corticosteroid treatment are not eligible for enrollment.
* Patients with psychiatric disorders, substance abuse, or social issues that affect compliance are not eligible for enrollment after physician review.
* Patients who are allergic to or contraindicated for PD-1 monoclonal antibodies, VEGF monoclonal antibodies, or chemotherapy drugs.

Withdrawl criteria:

* Incorrectly enrolled participants. Those who have not yet received treatment in this study should be immediately withdrawn, and their information will not be included in the study analysis. If treatment has already begun, the investigator should assess the participant's benefit-risk profile and then decide whether to withdraw. If withdrawal is necessary, the participant should exit the study after completing treatment and follow-up and will not be included in the efficacy analysis of this study, but must be included in the safety analysis.
* Participants who experience the following during the pre-treatment evaluation phase: new systemic diseases or worsening of existing systemic diseases that meet exclusion criteria; voluntary withdrawal, loss to follow-up, or death; poor compliance.
* Participants whom the investigator deems necessary to exclude. The investigator must report the reason for exclusion to the principal investigator and obtain consent. Those who have not yet received treatment in this study should be immediately withdrawn, and their information will not be included in the study analysis. If treatment has already begun, the participant should exit the study after completing treatment and follow-up and will not be included in the efficacy analysis of this study, but must be included in the safety analysis.
* Participants may request to withdraw from the clinical trial at any time during the trial process.
* Participants who experience serious adverse events during the trial, and whom the investigator deems should stop participating in the trial.
* Participants whose condition worsens during the trial, potentially threatening their life, or who develop other conditions that affect trial observations.
* Participants who are lost to follow-up or die during the treatment phase.
* Participants who use chemotherapy, traditional Chinese medicine, other immunotherapy drugs, radiotherapy sensitizers, or other agents that affect efficacy and toxicity evaluation during the trial period.
* Participants in whom serious deviations occur during the implementation of the clinical trial protocol, making it difficult to evaluate the drug's effect; those with poor compliance.

Exit criteria:

* Wrong enrollees who did not meet the inclusion criteria;
* Serious protocol violations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 1 year
  The time from the start of drug treatment until the documentation of disease progression or death from any cause, assessed according to the RECIST 1.1 criteria. Patients who are still alive at the time of analysis will have their last contact date used as the cutoff date.

SECONDARY OUTCOMES:
Overall Survival (OS) | 1 year
  The time from the start of drug treatment until death from any cause. Patients who are still alive at the time of analysis will have their last contact date used as the cutoff date.
Objective Response Rate (ORR) | 1 year
  The percentage of participants who achieve a Complete Response (CR) or Partial Response (PR) after treatment, assessed according to the RECIST 1.1 criteria.
Treatment-related adverse event (TRAE) | 1 year
  Investigator-assessed treatment-related adverse events were recorded and assessed according to CTCAE5.0.